CLINICAL TRIAL: NCT03930459
Title: Clinical Trial to Compare the Efficacy of Ex-situ Normothermic Perfusion With Cold Storage in the Transplant With Steatotic Liver Graft.
Brief Title: Efficacy of Ex-situ Normothermic Perfusion Versus Cold Storage in the Transplant With Steatotic Liver Graft.
Acronym: ORGANOXLAFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORGANOXLAFE
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2019-08

CONDITIONS: Liver Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static cold storage (SCS) (Experimental): Traditional method of organ preservation which involves flushing of cold preservation solution following complete dissection and interruption of blood supply to the donor organ. Although cold preservation slows metabolism by 10- to 12-fold, substantial anaerobic activity continues even at ice temperature. This lead to the generation of reactive oxygen species that are the basis of ischaemia-reperfusion injury, when the organ is re-exposed to oxygenated blood at the time of transplantation. This damage, exacerbated by any prior injury, limits the maximum safe preservation time of the donor organ.
  Interventions: Procedure: Static cold storage (SCS)
- Normothermic machine perfusion (NMP) (Experimental): The main goal of NMP is to optimize graft preservation by mimicking physiological conditions. The perfused organ is supplied with nutrients and oxygen to maintain metabolic hemostasis. Under these conditions, ATP and glycogen reserves can be maintained or actively restored. At the same time, toxic products from the cellular milieu are continuously eliminated, so the cell-mediated injury phase of reperfusion injury can be minimized. Thus, ischemic injury is avoided and the activation of cell death cascades is prevented. This allows both hepatocellular and biliary protection.
  Interventions: Device: Normothermic machine perfusion (NMP)

INTERVENTIONS:
Procedure: Static cold storage (SCS) — The liver is flushed and cooled with specialist preservation fluid, then stored in an icebox.
  Arms: Static cold storage (SCS)
Device: Normothermic machine perfusion (NMP) — During NMP, the liver is perfused with oxygenated blood, medications and nutrients at normal body temperature to maintain a physiological milieu.
  Arms: Normothermic machine perfusion (NMP)

SUMMARY:
Prospective, randomized, controlled clinical trial to determine the overall efficacy of normothermic machine perfusion (NMP) for steatotic liver preservation versus traditional static cold storage (SCS), in 50 liver transplant recipients with 1-year follow-up.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical trial comparing static cold storage (SCS) versus normothermic machine perfusion (NMP) for organ preservation before liver transplantation with steatotic livers (between 30 % and 60% of histologic macrovesicular steatosis), in order to:

Main Objective:

To compare the effect of NMP versus SCS in preventing preservation injury and graft dysfunction, as measured by highest transaminase levels during the first week after liver transplantation.

Secondary Objectives:

* To compare graft and patient survival between the NMP and SCS steatotic livers.
* To compare the liver biochemical function between the NMP and SCS steatotic livers.
* To compare the physiological response to the reperfusion between the NMP and SCS steatotic livers.
* To compare the evidence of reperfusion injury between the NMP and SCS steatotic livers.
* To compare the evidence of ischemic cholangiopathy between the NMP and SCS steatotic livers.

ELIGIBILITY:
Inclusion Criteria:

LIVER DONOR:

* Donors older than 16 years
* Liver donation grafts due to brain death
* Steatosis confirmed by histological study (between 30% and 60% of macrovesicular steatosis)

LIVER RECIPIENT:

* Adult patients (18 years or older)
* Active liver transplant waiting list candidate
* Able to give informed consent

Exclusion Criteria:

LIVER DONOR:

* Living donors
* Liver destined to the transplant "split"
* Donor age <16 years
* Donation after death due to asystole.
* When the biopsy establishes a steatosis ≥ 50%, patients who fulfill at least 3 of the following 5 risk factors will be excluded: Transaminases (AST and ALT) ≥ 200 U / L; Age ≥ 55 years; Hypernatremia ≥ 155 mEq / L; Cardiovascular risk factors, at least 2 of the following 5: DM, HTA, IMC ≥ 35, Active smoking, ischemic stroke; Days of stay in ICU ≥ 4 days with vasoactive drugs (noradrenaline or dobutamine at any dose)

LIVER RECIPIENT:

* Age under 18
* Acute/fulminant hepatic failure
* Transplant of more than one organ (for example, liver and kidney)
* Rejection of informed consent
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Peak of transaminases (AST and ALT) | Day 1 post-transplant.
Peak of transaminases (AST and ALT) | Day 3 post-transplant.
Peak of transaminases (AST and ALT) | Day 5 post-transplant.
Peak of transaminases (AST and ALT) l | Day 7 post-transplant.

SECONDARY OUTCOMES:
Primary graft failure | Day 10 post-transplant.
  Primary graft failure: irreversible graft dysfunction that requires emergency hepatic replacement during the first 10 days after liver transplantation, in the absence of technical or immunological causes.
Graft survival | Day 30 post-transplant, month 6 post-transplant, month 12 post-transplant.
Patient survival | Day 30 post-transplant, month 6 post-transplant, month 12 post-transplant.
Post-reperfusion syndrome, measured by mean arterial pressure (MAP) levels | During the first 5 minutes after reperfusion
  Post-reperfusion syndrome is defined as a decrease in mean arterial pressure (MAP) of more than 30% of the baseline value for more than one minute during the first five minutes after reperfusion. This will be evaluated in the context of the use of vasopressors.
Biochemical function of the liver measured by Bilirubin post-transplant levels | Day 1, day 3, day 5, day 7, day 30, month 6, month 12 post- transplant
Biochemical function of the liver measured by GGT post-transplant levels | Day 1, day 3, day 5, day 7, day 30, month 6, month 12 post- transplant
Biochemical function of the liver measured by AST post-transplant levels | Day 1, day 3, day 5, day 7, day 30, month 6, month 12 post- transplant
Biochemical function of the liver measured by ALT post-transplant levels | Day 1, day 3, day 5, day 7, day 30, month 6, month 12 post- transplant
Biochemical function of the liver measured by INR post-transplant levels | Day 1, day 3, day 5, day 7, day 30, month 6, month 12 post- transplant
Early graft dysfunction | 7 days post-transplant
  Defined by:
  1. Bilirubin > 10 mg / dl daily 7 after transplant
  2. INR > 1.6 on day 7 after transplantation.
  3. Peak AST and ALT > 2000 IU / L in the first 7 days after transplantation
Intensive care stay duration | Day 30
Hospital stay duration | Day 30
Renal replacement therapy need | Day 30, month 6, month 12 post- transplant
Intraoperative thromboelastogram result | In transplant surgery
Histological evidence of reperfusion injury | In transplant surgery
  Post-reperfusion biopsies will be compared with baseline pre-reperfusion biopsies and classified according to standard histological criteria (blind comparison to third parties).
Evidence of biliary stenosis in magnetic resonance cholangiography (MRS). | 6 months after transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

REFERENCES:
- [Background] Garcia-Valdecasas JC, Tabet J, Valero R, Taura P, Rull R, Garcia F, Montserrat E, Gonzalez FX, Ordi J, Beltran J, Lopez-Boado MA, Deulofeu R, Angas J, Cifuentes A, Visa J. Liver conditioning after cardiac arrest: the use of normothermic recirculation in an experimental animal model. Transpl Int. 1998;11(6):424-32. doi: 10.1007/s001470050169. PMID 9870271
- [Background] St Peter SD, Imber CJ, Lopez I, Hughes D, Friend PJ. Extended preservation of non-heart-beating donor livers with normothermic machine perfusion. Br J Surg. 2002 May;89(5):609-16. doi: 10.1046/j.1365-2168.2002.02052.x. PMID 11972552
- [Background] Imber CJ, St Peter SD, Lopez de Cenarruzabeitia I, Pigott D, James T, Taylor R, McGuire J, Hughes D, Butler A, Rees M, Friend PJ. Advantages of normothermic perfusion over cold storage in liver preservation. Transplantation. 2002 Mar 15;73(5):701-9. doi: 10.1097/00007890-200203150-00008. PMID 11907414
- [Background] Gaffey MJ, Boyd JC, Traweek ST, Ali MA, Rezeig M, Caldwell SH, Iezzoni JC, McCullough C, Stevenson WC, Khuroo S, Nezamuddin N, Ishitani MB, Pruett TL. Predictive value of intraoperative biopsies and liver function tests for preservation injury in orthotopic liver transplantation. Hepatology. 1997 Jan;25(1):184-9. doi: 10.1002/hep.510250134. PMID 8985288
- [Background] Karayalcin K, Mirza DF, Harrison RF, Da Silva RF, Hubscher SG, Mayer AD, Buckels JA, McMaster P. The role of dynamic and morphological studies in the assessment of potential liver donors. Transplantation. 1994 May 15;57(9):1323-7. doi: 10.1097/00007890-199405150-00006. PMID 8184469
- [Background] Abraham S, Furth EE. Quantitative evaluation of histological features in "time-zero" liver allograft biopsies as predictors of rejection or graft failure: receiver-operating characteristic analysis application. Hum Pathol. 1996 Oct;27(10):1077-84. doi: 10.1016/s0046-8177(96)90287-7. PMID 8892594
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Background] Chung IS, Kim HY, Shin YH, Ko JS, Gwak MS, Sim WS, Kim GS, Lee SK. Incidence and predictors of post-reperfusion syndrome in living donor liver transplantation. Clin Transplant. 2012 Jul-Aug;26(4):539-43. doi: 10.1111/j.1399-0012.2011.01568.x. Epub 2011 Dec 14. PMID 22168355
- [Background] Hilmi I, Horton CN, Planinsic RM, Sakai T, Nicolau-Raducu R, Damian D, Gligor S, Marcos A. The impact of postreperfusion syndrome on short-term patient and liver allograft outcome in patients undergoing orthotopic liver transplantation. Liver Transpl. 2008 Apr;14(4):504-8. doi: 10.1002/lt.21381. PMID 18383079
- [Background] Glanemann M, Langrehr JM, Stange BJ, Neumann U, Settmacher U, Steinmuller T, Neuhaus P. Clinical implications of hepatic preservation injury after adult liver transplantation. Am J Transplant. 2003 Aug;3(8):1003-9. doi: 10.1034/j.1600-6143.2003.00167.x. PMID 12859537
- [Background] Eisenbach C, Encke J, Merle U, Gotthardt D, Weiss KH, Schneider L, Latanowicz S, Spiegel M, Engelmann G, Stremmel W, Buchler MW, Schmidt J, Weigand MA, Sauer P. An early increase in gamma glutamyltranspeptidase and low aspartate aminotransferase peak values are associated with superior outcomes after orthotopic liver transplantation. Transplant Proc. 2009 Jun;41(5):1727-30. doi: 10.1016/j.transproceed.2009.01.084. PMID 19545716
- [Background] Nasralla D, Coussios CC, Mergental H, Akhtar MZ, Butler AJ, Ceresa CDL, Chiocchia V, Dutton SJ, Garcia-Valdecasas JC, Heaton N, Imber C, Jassem W, Jochmans I, Karani J, Knight SR, Kocabayoglu P, Malago M, Mirza D, Morris PJ, Pallan A, Paul A, Pavel M, Perera MTPR, Pirenne J, Ravikumar R, Russell L, Upponi S, Watson CJE, Weissenbacher A, Ploeg RJ, Friend PJ; Consortium for Organ Preservation in Europe. A randomized trial of normothermic preservation in liver transplantation. Nature. 2018 May;557(7703):50-56. doi: 10.1038/s41586-018-0047-9. Epub 2018 Apr 18. PMID 29670285